CLINICAL TRIAL: NCT03430258
Title: High-flow Nasal Cannula Oxygen Therapy With the Chest Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19850703
Record Dates: First submitted 2018-01-04; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Blunt Thoracic Injury; Lung Ultrasound Score

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional oxygen therapy (Placebo Comparator): oxygen was delivered by a nasal cannula or nonrebreather mask
  Interventions: Device: Conventional oxygen therapy
- High-flow Nasal Cannula Oxygen Therapy (Active Comparator): High-flow Nasal Cannula Oxygen Therapy
  Interventions: Device: high-flow nasal cannula

INTERVENTIONS:
Device: high-flow nasal cannula — high flow of air with supplemental oxygen was delivered by an Optiflow cannula interface using an AIRVO 2 blower humidifier
  Arms: High-flow Nasal Cannula Oxygen Therapy
Device: Conventional oxygen therapy — Conventional oxygen therapy
  Arms: conventional oxygen therapy

SUMMARY:
This prospective randomized controlled study was conducted in the emergency intensive care units (EICU) of the second affiliated hospital Zhejiang university school of medicine, a large tertiary university hospital in HangZhou, China.The aim of this randomized study was to compare the effectiveness of high-flow nasal cannula with conventional oxygen therapy in ICU patients with blunt thoracic injury.

DETAILED DESCRIPTION:
This prospective randomized controlled study was conducted in the emergency intensive care units (EICU) of the second affiliated hospital Zhejiang university school of medicine, a large tertiary university hospital in HangZhou, China.The aim of this randomized study was to compare the effectiveness of high-flow nasal cannula with conventional oxygen therapy in ICU patients with blunt thoracic injury.

ELIGIBILITY:
Inclusion Criteria:

- The trauma registry was used to identify patients with moderate to severe blunt thoracic injury (abbreviated injury scale (AIS) chest score ≥3) admitted to the ICU

Exclusion Criteria:

1. had intubation and used the mechanical ventilation within 2 hours
2. had the emergency surgerys within 2 hours
3. patients can not accessed by transthoracic lung ultrasound because of the sever aerodermectasia or pneumothorax
4. the Glasgow Coma Scale <8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
compare the effectiveness of high-flow nasal cannula with conventional oxygen therapy in ICU patients with blunt thoracic injury. | 72 hours
  High-flow nasal cannula could reduce the intube rate of patients with blunt thoracic injury,and improve the the lung aeration for patients with thoracic injury

SECONDARY OUTCOMES:
number of days in ICU | 7 days
  High-flow nasal cannula could reduce the number of days for the patients treatments in ICU

IPD SHARING:
Plan to Share IPD: No